CLINICAL TRIAL: NCT07085624
Title: Early Optimization of Ceftazidime Regimen in Critical Care
Acronym: FORTOPTIM_1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Direction Générale de l'Offre de Soins (Other Government); GIRCI Auvergne Rhône-Alpes (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24PH176_1; 2024-519783-41-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-25; First posted 2025-07-25 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Infection in ICU; Sepsis; Septic Shock; Pseudomonas Aeruginosa Infection
Keywords: ceftazidime; intensive care unit; pharmacokinetics; individualised dosing regimen
MeSH Terms: conditions — Sepsis; Shock, Septic; Pseudomonas Infections | interventions — Ceftazidime

STUDY DESIGN:
Intervention Model Description: Randomization comparing 2 therapeutic strategies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ceftazidime standard dosage regimen (Active Comparator): Loading dose 2g
  Maintenance dose :
  6g/d if GFR (Glomerular Filtration Rate) ≥ 60 3g/d if GFR between 30 and 60 1.5g/d if GFR between 15 and 30
  Interventions: Drug: ceftazidime; Biological: plasma ceftazidime dosage
- ceftazidime optimised dosage regimen (Experimental): Loading dose 4g
  Maintenance dose :
  6g/d if GFR (Glomerular Filtration Rate) ≥ 60 3g/d if GFR between 30 and 60 1.5g/d if GFR between 15 and 30
  Interventions: Drug: ceftazidime; Biological: plasma ceftazidime dosage

INTERVENTIONS:
Drug: ceftazidime — ceftazidime loading dose and maintenance dose
Biological: plasma ceftazidime dosage — plasma ceftazidime dosage kinetics will be performed according to an optimal D- sampling plan (4 measurements per subject: T0+5min, T0+3h, T0+6h, T0+24h, PFIM software).
  T0 corresponds to the time to administer the ceftazidime loading dose.

SUMMARY:
Hospital-acquired infections, most of which are caused by Gram-negative bacteria, are common in intensive care units and have a major impact on patient prognosis. Patient survival in severe sepsis and septic shock depends on the early administration of appropriate antibiotic therapy, with mortality increasing by 7.6% for each hour of delay, justifying the probabilistic use of broad-spectrum antibiotics such as ceftazidime, an essential betalactamine, particularly used for its activity against Pseudomonas aeruginosa, a frequent pathogen in nosocomial infections.

It is currently recommended that ceftazidime should initially be administered as a 2g loading dose, followed by maintenance treatment by continuous infusion, at a dose adapted to renal function.

The recommended dosage regimen, with its 2g loading dose, was developed using the median value of parameters from a pharmacokinetic model. This explains the findings of many critical care studies, which have found that 40-60% of patients initially have concentrations below target with the recommended dosing regimen.

In the context of critical care, maintaining concentrations within the target therapeutic range is difficult due to variations in the elimination clearance of ceftazidime. Ceftazidime is mainly eliminated by the kidneys. Critical patients may have increased glomerular filtration rate, or, conversely, impaired renal function, with rapid variations in the event of severe infection. This leads to high intra- and inter-individual variability, and increases the risk of antibiotic under- or overdose when the maintenance dose is administered at a fixed dose (6g/d continuously). This high variability can also be observed in the volume of distribution (capillary leakage, oedema, perfusion volumes, effusions ...).

In order to propose an individualised dosing regimen, we therefore propose an iterative randomised study to :

* Step 1: FORTOPTIM_1 Evaluation of an optimised dosage regimen based on literature data compared with the standard psological regimen.
* Step 2: FORTOPTIM_2 Build a pharmacokinetic model from the prospective data obtained in step 1. Based on this model, an individualised dosage regimen (loading dose and maintenance dose) will be obtained for step 3.
* Step 3: FORTOPTIM_3 Prospectively evaluate in a randomised trial the individualised dosing regimen previously defined (Step 2) by comparing it to the best dosing regimen determined in Step 1 or to the standard dosing regimen if there is no significant difference in Step 1.

ELIGIBILITY:
Inclusionn criteria:

* Patient hospitalized in intensive care unit for an expected duration of at least 72 hours, with an infection for which initiation of ceftazidime therapy is being considered.
* Patient with an arterial catheter for blood sampling.
* Patients affiliated to or entitled under a social security scheme.

Exclusion Criteria:

* Pregnant woman, parturient, nursing mother;
* Person deprived of liberty, hospitalized without consent,
* Adults under legal protection (guardianship-curatorship)
* Patients undergoing extra-renal purification or whose CKD-EPI at the start of treatment is less than 15 ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with a ceftazidime concentration equal to or above the target concentration threshold (35 mg/L) at both 3h and 24h after the first administration, and below the toxicity threshold of 100 mg/L. | 24 hours

SECONDARY OUTCOMES:
Patient severity assessed using the SOFA (Sequential Organ Failure Assessment Score) | day 7
  SOFA score from 0 to 24 The higher the score (24), the greater the incidence of organ failure
death | day 28
Occurrence of neurological adverse events defined as: seizure, myoclonus, encephalopathy or delirium, altered consciousness (Glasgow score) | day 28
Occurrence of an overdose defined as a concentration greater than 100 mg/L. | day 28
Renal function assessment | day 28
  creatinine clearance (mL/mn) with the CKD-EPI (Chronic Kidney Disease - Epidemiology Collaboration) equation
Time to reach PK/PD (pharmacokinetics/pharmacodynamics) targets | 24 hours

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CHU GRENOBLE, Médecine intensive, Grenoble
  - HCL Croix Rousse, Médecine intensive réanimation, Lyon
  - HCL Hôpital Edouard Herriot, Médecine intensive et réanimation, Lyon
  - CHU Nord, Médecine intensive et réanimation, Marseille
  - HCL Hôpital Lyon Sud, Médecine intensive réanimation, Pierre-Bénite
  - CHU ST-ETIENNE - Médeine Intensive Réanimation, Saint-Etienne
  - CHU ST-ETIENNE, Médecine intensive Réanimation B, Saint-Etienne
  - CHU ST-ETIENNE, Réanimation Néphrologie, Saint-Etienne